CLINICAL TRIAL: NCT02554201
Title: Efficacy of Electrical Pudendal Nerve Stimulation for Neurogenic Lower Urinary Tract Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Institute of Acupuncture, Moxibustion and Meridian (Other)
Collaborators: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZYY201501
Record Dates: First submitted 2015-08-24; First posted 2015-09-18 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Spinal Cord Injuries; Lower Urinary Tract Symptoms; Dysuria; Incontinence
Keywords: pudendal nerve modulation; transanal/transvaginal electrical stimulation
MeSH Terms: conditions — Spinal Cord Injuries; Lower Urinary Tract Symptoms; Dysuria

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Electrical pudendal nerve stimulation (Experimental): Electrical pudendal nerve stimulation At a frequency of 2.0 Hz and a moderate intensity (25~35 mA); 60 minutes three times a week for a total of four weeks
  Interventions: Device: Electrical pudendal nerve stimulation
- Transvaginal electrical stimulation (Active Comparator): At a current intensity of < 60 mA (as high as possible to get a contraction) and frequencies of 15 Hz and 85 Hz (alternate 3-min periods of stimulation); 30 min three times a week for a total of four weeks.
  Interventions: Device: Transvaginal electrical stimulation

INTERVENTIONS:
Device: Electrical pudendal nerve stimulation — Four sacral points are selected. The two upper points are located about 1 cm bilateral to the sacrococcygeal joint. Needles of 0.40 Х 100 mm are inserted perpendicularly to the upper points to a depth of 80 to 90 mm to produce a sensation referred to the urethra or the anus. The two lower points are about 1 cm bilateral to the tip of the coccyx. Needles of 0.40 Х 100 or 125 mm are inserted obliquely to the lower points towards the ischiorectal fossa to a depth of 90 to 110 mm to produce a sensation referred to the urethra. After the sensation referred to the above regions is produced, each of two pairs of electrodes from a G6805-2 Multi-Purpose Health Device is connected with the two ipsilaterally needles.
  Arms: Electrical pudendal nerve stimulation
Device: Transvaginal electrical stimulation — A neuromuscular stimulation therapy system (PHENIX USB 4，Electronic Concept Lignon Innovation, France) is used for TES
  Arms: Transvaginal electrical stimulation

SUMMARY:
The main goal to treat early NLUTS is to relieve lower urinary tract syndrome and prevent from late complications. The present study is to evaluate the efficacy of electrical pudendal nerve stimulation (EPNS) and transanal/transvaginal electrical stimulation (TES) in NLUTD.The study design consists of a non-randomized, parallel controlled trial. A total of 60 eligible patients will be involved and divided into EPNS or TES group according to their location of medical treatment. The primary endpoint is lower urinary tract syndromes (ICIQ-FLUTS/MLUTS). The second endpoint is assessment of daily life Qol (ICIQ-LUTSqol), and residual urine volume.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+ years;
* Diagnosed as NLUTD;
* Incomplete spinal cord injury (SCI), including but not limited to conus medullaris syndrome, cauda equina syndrome, etc.;
* Radical pelvic surgery: including but not limited to total hysterectomy etc.;
* Informed consent signed.

Exclusion Criteria:

* Anatomical bladder outlet obstruction (e.g., prostate enlargement, tumors);
* NLUTD induced by stroke, multiple sclerosis, HIV, diabetes mellitus, drug, and inflammation or tumor of central nervous system etc.;
* Lower urinary tract infections;
* Unwillingness to participate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
A questionaire to measure the severity of lower urinary tract symptoms (male/female) | 1.5 years

SECONDARY OUTCOMES:
A questionaire to evaluate the Qol | 1.5 years
Residual urine volume | 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Siyou Wang, Master, Study Chair — Shanghai research institute of acupuncture and meridian
Locations (1):
- Shanghai research institute of acupuncture and meridian, Shanghai, China